CLINICAL TRIAL: NCT00725465
Title: Prospective Evaluation of Combined Laparoscopy With CO2 Intraoperative Colonoscopy Treatment for Colorectal Lesions
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0411007608
Record Dates: First submitted 2008-07-24; First posted 2008-07-30 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Polyps
Keywords: laparoscopy; CO2 colonoscopy; intraoperative CO2 colonoscopy; combined Lap-CO2 procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAP surgery with CO2 colonoscopy: 30 surgical patients, male and female undergoing laparoscopic surgical treatment for colorectal conditions such as neoplasm or rectal prolapse managed with intra-operative carbon dioxide (co2)colonoscopy for standard care of their medical condition.

SUMMARY:
The purpose of this study is to evaluate prospectively the usefulness of IC-CO2(intraoperative colonoscopy (IC) using carbon dioxide (CO2)) in colon and rectal surgical practice, coincident with laparoscopic surgery, and assess whether it provides useful information that influences the type of surgical therapy intended. Investigators will further define the safety and extent of bowel distension when using IC-CO2.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate prospectively the usefulness of IC-CO2(intraoperative colonoscopy (IC) using carbon dioxide (CO2)) in colon and rectal surgical practice, coincident with laparoscopic surgery, and assess whether it provides useful information that influences the type of surgical therapy intended. Investigators will further define the safety and extent of bowel distension when using IC-CO2. Furthermore, the investigators will evaluate the therapy and technique of using this combined approach to the treatment of colorectal polyps and other localized, benign lesions of the large intestine. In this study, the colonoscope is used both as a diagnostic and therapeutic tool, and is often used in order to avoid a major bowel resection, yet effectively treat localized lesions of the large intestine.

The hypothesis of this study is that IC-CO2 will provide useful information which does affect surgical decision making at the time of operation, and that it is safe and does not result in any significant bowel distention during or immediately after the procedure. We additionally hypothesize that certain localized lesions of the intestines may be treated using a combined laparoscopic-IC-CO2 approach to effectively treat the underlying disease, minimize risks to the patient, and avoid a major bowel resection.

ELIGIBILITY:
Inclusion Criteria:

* All patients (male and female) greater than 18 years of age who undergo a laparoscopic surgical procedure that utilizes intra-operative colonoscopy will be approached to participate in this study

Exclusion Criteria:

* Patients under 18 year of age
* Patients with severe Renal Diseases
* Ascites
* COPD (severe)
* Liver insufficiency (severe) with coagulopathy
* Dialysis
* Sleep Apnea
* Patient pregnant
* Multiple previous surgeries
* Subject is incapable of understanding the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 surgical patients, male and female undergoing laparoscopic surgical treatment for colorectal conditions such as neoplasm or rectal prolapse managed with intra-operative carbon dioxide (co2)colonoscopy for standard care of their medical condition. Multiple measurments of Arterial Blood Gass will be performed and evaluated.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
arterial blood gas (ABG) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Milsom, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College, New York, New York, United States

REFERENCES:
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/21607827